CLINICAL TRIAL: NCT07341282
Title: Investigation of Vancomycin Efficacy in Patients With Ulcerative Colitis and Primary Sclerosing Cholangitis
Acronym: DRIVE-UP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Weston Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRIVE_UP2025
Record Dates: First submitted 2025-12-02; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC); Primary Sclerosing Cholangitis (PSC)
Keywords: Ulcerative Colitis; Primary Sclerosing Cholangitis; Vancomycin; Randomized Control Trial
MeSH Terms: conditions — Colitis, Ulcerative; Cholangitis, Sclerosing | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Participants will:
  Be randomized to receive either vancomycin or placebo orally twice daily for 4 weeks.
  Undergo clinical assessments including Mayo scoring, endoscopic evaluation, and laboratory testing at baseline, week 4, and follow-up.
  After 4 weeks, have the option to receive open-label vancomycin for an additional 4 weeks.
  Provide stool and blood samples for microbiome and biochemical analyses.
  Be monitored for adverse events and treatment adherence throughout the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): 4 weeks blinded placebo followed by optional 4 weeks open-label vancomycin.
  Interventions: Drug: Placebo (blinded); Drug: Vancomycin (open-label extension)
- Vancomycin (Experimental): 4 weeks blinded oral vancomycin followed by optional additional 4 weeks open-label vancomycin.
  Interventions: Drug: Vancomycin (blinded); Drug: Vancomycin (open-label extension)

INTERVENTIONS:
Drug: Placebo (blinded) — Identical placebo capsule administered orally twice daily for 4 weeks.
  Arms: Placebo Comparator
Drug: Vancomycin (blinded) — Vancomycin 250 mg administered orally twice daily for 4 weeks.
  Arms: Vancomycin
Drug: Vancomycin (open-label extension) — Vancomycin 250 mg administered orally twice daily for 4 weeks (optional extension offered to both arms).

SUMMARY:
This clinical trial tests if oral vancomycin can safely treat active ulcerative colitis (UC) in adults who also have primary sclerosing cholangitis (PSC), a liver condition. The main questions it aims to answer are:

* Can oral vancomycin improve UC symptoms as measured by Mayo score at 4 weeks?
* Is oral vancomycin safe and tolerable in this patient group?

Participants will be compared to see if vancomycin works better than placebo. Participants will:

* Take oral vancomycin (250 mg twice daily) or identical placebo capsules for 4 weeks
* Have the option for 4 more weeks of open-label vancomycin after the blinded phase
* Attend clinic visits at baseline, week 4, and follow-up for Mayo scoring, endoscopy, blood/stool tests, and safety checks
* Track treatment adherence and side effects

The study primarily assesses if the trial can recruit 14 participants, retain them, achieve good adherence, and follow protocol procedures (feasibility). Secondary goals include safety (adverse events) and early signs of benefit in UC activity, liver tests, and gut bacteria balance. This pilot will guide larger future studies.

DETAILED DESCRIPTION:
This is an investigator-initiated feasibility study designed to rigorously characterize clinical response signals, safety parameters, and feasibility metrics in adults with co-existing PSC and UC, a population where microbiome-targeted immune modulation is hypothesized to influence disease activity.

Randomization & Allocation Governance

* Randomization will be implemented using validated computer-generated randomization software, with the allocation sequence generated by a study statistician not involved in clinical assessments.
* Allocation concealment will be maintained through centralized pharmacy control. An independent pharmacist will assign treatment codes and release sequentially numbered study medication containers.
* Blinding integrity will be preserved through visual and packaging equivalence, sequential drug accountability logs, and restricted access to treatment codes until database lock.
* Emergency unblinding is permitted only when required for clinical management, and all unblinding events will be documented, timestamped, and reviewed by the DSMC.

Clinical Visit & Assessment Schedule

Participants will complete a structured study visit pathway:

* Screening (≤14 days before baseline): medical history review, infection risk screening, liver disease stability assessment, and confirmation of clinical trial eligibility documentation.
* Baseline (Week 0): clinical evaluation, safety labs, medication reconciliation, and flexible sigmoidoscopy performed by credentialed endoscopists using a standardized endoscopic scoring handbook.
* Week 2 & 4: in-clinic evaluation, adverse event review, safety labs, and compliance verification via pill count and participant diary reconciliation.
* Week 8 (extension follow-up): final safety labs, medication reconciliation, delayed adverse event capture, and optional qualitative feasibility interview.

Adherence & Safety Surveillance

* Participants will complete weekly digital symptom and adherence diaries capturing stool frequency, rectal bleeding trends, abdominal pain patterns, and missed doses.
* Safety labs include CBC, creatinine, liver panel, CRP, albumin, electrolytes, and will be evaluated at baseline, week 2, 4, and 8.
* A hepatologist co-investigator will review liver safety signals in real-time, given PSC-specific vulnerability to hepatic decompensation.
* Audiology risk is screened at entry, and any symptoms concerning for ototoxicity will prompt same-week clinical review.

Data Capture & Monitoring Integrity

* All data will be captured in a secure Excel file
* Endoscopic images will be stored in a secured institutional imaging server.
* A pre-registered statistical analysis plan will be finalized before unblinding, with analysis scripts locked prior to treatment code release.

Safety Governance Structure

The DSMC will provide independent oversight and safety adjudication:

* Quarterly DSMC meetings will evaluate cumulative safety logs, recruitment feasibility, protocol deviations, and unblinding reports.
* A real-time SAE notification system ensures DSMC alert within 24 hours of serious adverse event reporting.
* Pre-defined individual, arm-level, and whole-trial safety review thresholds are codified in the DSMC governance charter to support early pause or protocol modification when required.

Regulatory & Ethical Compliance

The trial will follow all institutional and international regulatory standards:

* ICH-GCP
* Institutional Research Ethics Board approval
* DSMC governance charter
* GMP-aligned pharmacy accountability procedures

ELIGIBILITY:
Inclusion Criteria

* Adults aged ≥18 years.
* Confirmed diagnosis of UC and PSC.
* Moderate to severe UC disease activity (total Mayo score ≥5; endoscopic subscore ≥2).
* Informed consent provided. Exclusion Criteria
* Diagnosis of Crohn's disease or indeterminate colitis.
* Fulminant colitis or need for immediate surgical intervention.
* Use of antibiotics or probiotics within the past 4 weeks (for microbiome substudy).
* Decompensated liver disease (Child-Pugh B/C).
* Severe Renal Impairment (CrCl <30mL/min)
* Active untreated infection.
* Pregnancy or lactation.
* Prior allergy or intolerance to Vancomycin
* History of hearing loss or current hearing problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  Proportion of eligible participants who provide consent and are enrolled in the study (number enrolled ÷ number eligible approached), with a target of 14 participants within 12 months.
Retention rate | 12 months
  Proportion of enrolled participants who complete all protocol-specified study visits and assessments at 12 months (number completing all follow-up visits ÷ number enrolled).
Treatment adherence | 12 months
  Proportion of prescribed oral vancomycin doses taken over the treatment period, assessed by pill counts and/or medication diary (number of doses taken ÷ number of doses prescribed).
Protocol compliance with study procedures | 12 months
  Proportion of participants with all required visits, laboratory tests, and assessments completed per protocol (number fully compliant ÷ number enrolled); may also include rate of major protocol deviations.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | 12 months
  Proportion of participants with at least one treatment-emergent adverse event (AE) or serious adverse event (SAE)
Severity and type of adverse events | 12 months
  Number of treatment-emergent AEs and SAEs by maximum severity grade (mild/moderate/severe) and type (MedDRA preferred term).
Relationship of adverse events to oral vancomycin | 12 months
  Proportion of AEs/SAEs assessed by investigator as related to intervention (number related ÷ total events).
Patient-reported tolerability of oral vancomycin | 12 months
  Mean score of side effect frequency and impact on 0-10 scale (0=no impact, 10=worst impact) via study questionnaire.

OTHER OUTCOMES:
Exploratory Endpoints (Change in Mayo Score from baseline) | 12 months
  Change in partial Mayo Clinic Score (range 0-12 points, higher scores indicate greater ulcerative colitis disease activity) from baseline to 12 months.
Exploratory Endpoints (Change in serum liver enzymes from baseline) | 12 months
  Change in serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels (units: U/L) from baseline to 12 months.
Exploratory Endpoints (Change in gut microbiome diversity from baseline) | 12 months
  Change in gut microbiome diversity (Shannon index, unitless) measured by 16S rRNA sequencing of fecal samples from baseline to 12 months.
Exploratory Endpoints (Change in fecal bile acids from baseline) | 12 months
  Change in total fecal bile acid concentration (units: μmol/g) measured by mass spectrometry from baseline to 12 months.
Exploratory Endpoints (Change in fecal short chain fatty acids from baseline) | 12 months
  Change in total fecal short chain fatty acid concentration (units: μmol/g), including acetate, propionate, and butyrate, measured by gas chromatography from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Narula, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital - Digestive Diseases Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data sharing policies would follow institutional and regulatory standards on data confidentiality and sharing.
  De-identified data shared upon request to qualified researchers with appropriate data use agreements, respecting participant confidentiality and ethical approvals.
  Patient demographics, primary data and data analysis can be shared.
Supporting Information: Study Protocol
Time Frame: Start Date is estimated in January 2026 - end date is estimated in December 2026.
Access Criteria: Access to IPD and supporting study documents will generally limited to qualified researchers who submit a reasonable scientific request and have the necessary expertise.
  The data shared would be de-identified or anonymized to protect participant confidentiality.
  Researchers might be granted access under data use agreements that specify the terms of use, including restrictions on re-identification and further sharing.
  Access is often facilitated through secure data repositories or by request through the trial sponsor or coordinating research unit after review and approval of the request.

REFERENCES:
- [Background] Arbabzada N, Dennett L, Meng G, Peerani F. The Effectiveness of Oral Vancomycin on Inflammatory Bowel Disease in Patients With Primary Sclerosing Cholangitis: A Systematic Review. Inflamm Bowel Dis. 2025 Jul 7;31(7):2027-2035. doi: 10.1093/ibd/izae257. PMID 39495039
- [Background] Shah A, Macdonald GA, Morrison M, Holtmann G. Targeting the Gut Microbiome as a Treatment for Primary Sclerosing Cholangitis: A Conceptional Framework. Am J Gastroenterol. 2020 Jun;115(6):814-822. doi: 10.14309/ajg.0000000000000604. PMID 32250997
- [Background] Al Sulais E, AlAmeel T, Alenzi M, Shehab M, AlMutairdi A, Al-Bawardy B. Colorectal Neoplasia in Inflammatory Bowel Disease. Cancers (Basel). 2025 Feb 16;17(4):665. doi: 10.3390/cancers17040665. PMID 40002259
- [Background] Castano-Milla C, Chaparro M, Gisbert JP. Systematic review with meta-analysis: the declining risk of colorectal cancer in ulcerative colitis. Aliment Pharmacol Ther. 2014 Apr;39(7):645-59. doi: 10.1111/apt.12651. PMID 24612141
- [Background] Lutgens MW, van Oijen MG, van der Heijden GJ, Vleggaar FP, Siersema PD, Oldenburg B. Declining risk of colorectal cancer in inflammatory bowel disease: an updated meta-analysis of population-based cohort studies. Inflamm Bowel Dis. 2013 Mar-Apr;19(4):789-99. doi: 10.1097/MIB.0b013e31828029c0. PMID 23448792
- [Background] Lundberg Bave A, Bergquist A, Bottai M, Warnqvist A, von Seth E, Nordenvall C. Increased risk of cancer in patients with primary sclerosing cholangitis. Hepatol Int. 2021 Oct;15(5):1174-1182. doi: 10.1007/s12072-021-10214-6. Epub 2021 Aug 6. PMID 34357546
- [Background] Risques RA, Lai LA, Himmetoglu C, Ebaee A, Li L, Feng Z, Bronner MP, Al-Lahham B, Kowdley KV, Lindor KD, Rabinovitch PS, Brentnall TA. Ulcerative colitis-associated colorectal cancer arises in a field of short telomeres, senescence, and inflammation. Cancer Res. 2011 Mar 1;71(5):1669-79. doi: 10.1158/0008-5472.CAN-10-1966. PMID 21363920
- [Background] Ullman TA, Itzkowitz SH. Intestinal inflammation and cancer. Gastroenterology. 2011 May;140(6):1807-16. doi: 10.1053/j.gastro.2011.01.057. PMID 21530747
- [Background] Uzdzicki AW, Wawrzynowicz-Syczewska M. Characteristic features of ulcerative colitis with concomitant primary sclerosing cholangitis. Prz Gastroenterol. 2021;16(3):184-187. doi: 10.5114/pg.2021.108983. Epub 2021 Sep 17. PMID 34584578